CLINICAL TRIAL: NCT01066520
Title: A Randomized, Controlled, Multi-center Study on the Effectiveness of Traumeel S (Both Ointment and Gel) in Terms of Pain and Function Compared With a Topical NSAID in Athletes With Acute Ankle Sprain
Brief Title: TAASS-Traumeel Ointment and Gel Compared With a Topical NSAID in Athletes With Acute Ankle Sprain
Acronym: TAASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRS-ESP; 2008-007939-41 (EudraCT Number)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Sprain of Ankle
Keywords: ankle sprain; traumeel; diclofenac; antiinflammatory; time to normal function
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traumeel S ointment (Experimental): Traumeel S ointment 2 g, 3 times daily topical during 14 days
  Interventions: Drug: Traumeel S ointment
- Traumeel S gel (Experimental): Traumeel S gel 2 g, 3 times daily topical during 14 days
  Interventions: Drug: Traumeel S gel
- Diclofenac gel (Active Comparator): Diclofenac gel 2 g, 3 times daily topical during 14 days
  Interventions: Drug: Diclofenac gel

INTERVENTIONS:
Drug: Traumeel S ointment — 2 g, 3 times daily topical during 14 days
  Other Names: Traumeel S ointment, Traumeel S gel, Diclofenac gel
  Arms: Traumeel S ointment
Drug: Traumeel S gel — 2 g, 3 times daily topical during 14 days
  Arms: Traumeel S gel
Drug: Diclofenac gel — 2 g, 3 times daily topical during 14 days
  Arms: Diclofenac gel

SUMMARY:
The objective of this study is to determine the efficacy of Traumeel S (both ointment and gel) compared to another antiinflammatory drug called Diclofenac in patients with a sprained ankle.

DETAILED DESCRIPTION:
Study objective is the confirmatory proof of efficacy for Traumeel® S topical treatment, both ointment and gel, as compared to diclofenac topical treatment for patients with ankle sprain. In addition tolerability/safety of both drug preparations is to be compared, so that the benefit-risk relation can be determined.

ELIGIBILITY:
Inclusion criteria:

* Athletes with an acute unilateral ankle sprain of the lateral ligaments of the ankle joint both male and female
* Moderate (30-60 mm) to severe (>60 mm) pain according to the patient's assessment of ankle pain visual analogue scale (VAS) on weight bearing, unable to perform normal training / sports activities
* 18 - 40 years of age
* injury occurred within 24 hours of the first dose of study medication
* Willing and able to give written informed consent
* Available for the duration of the study

Exclusion Criteria:

* Similar injury affecting the same joint within the past 6 months
* bilateral ankle injury
* bed rest, hospitalization, surgery use of a non-removable rigid cast
* Clinically important abnormality for screening laboratory tests
* Debilitating acute or chronic illness
* Use of corticosteroids in the previous 8 weeks, any analgesics in the previous 6 hours, or 24 hours in case of long-acting NSAID, COX-2 specific inhibitors, or tramadol
* History of sensitivity to any component of the study drugs
* Unwilling or unable to comply with all the requirements of the protocol
* Participation in other studies within 4 weeks prior to study entry and or during the study participation
* Current substance or alcohol abuse that in the opinion of the investigator would interfere with compliance or with interpretation of the study result

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 449 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gonzalez de Vega, MD, Study Chair — National Coordinating Investigator
Locations (1):
- MEDYR Medicina Deportiva y Rehabilitación, Madrid, Spain

REFERENCES:
- [Derived] Gonzalez de Vega C, Speed C, Wolfarth B, Gonzalez J. Traumeel vs. diclofenac for reducing pain and improving ankle mobility after acute ankle sprain: a multicentre, randomised, blinded, controlled and non-inferiority trial. Int J Clin Pract. 2013 Oct;67(10):979-89. doi: 10.1111/ijcp.12219. Epub 2013 Jul 25. PMID 23889885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initiation date stage I(299 patients):24.08.2009, completion date stage I: 19.01.2011 Initiation date stage II(150 patients): 04.03.2011, completion date stage II: 12.09.2011 The evaluation criteria have not been changed in the different stages. The interim analysis after Stage I re-confirmed the originally calculated sample size.
Pre-assignment Details: Athletes of both sexes with acute unilateral sprain of the lateral ankle joint; 18 to 40 years of age; injury occurred within 24 hours of the first dose of study medication, with moderate (30-60mm) to severe (>60mm) pain on weight bearing.420 of the enrolled 449 patients have been selected into the ITT population. 447 patients received treatment
Groups:
- Traumeel S Ointment: Traumeel® S ointment, 2 g of ointment three times daily for 14 days, to sufficiently cover the area of the lesion, gently rubbing
- Traumeel S Gel: Traumeel® S gel, 2 g of gel three times daily for 14 days, to sufficiently cover the area of the lesion, gently rubbing
- Diclofenac Gel: NSAID gel (Diclofenac 1%; standard brand), 2 g of gel three times daily for 14 days, to sufficiently cover the area of the lesion, gently rubbing
Period: Overall Study
Arm/Group | Traumeel S Ointment | Traumeel S Gel | Diclofenac Gel
Started | 143 | 140 | 137
Completed | 143 | 140 | 137
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analyzed ITT population
Groups:
- Traumeel S Ointment: Traumeel S Ointment 2g, 3 times daily topical during 14 days
- Traumeel S Gel: Traumeel S Gel 2g, 3 times daily topical during 14 days
- Diclofenac Gel: Diclofenac Gel 2g, 3 times daily topical during 14 days
- Total: Total of all reporting groups
Arm/Group | Traumeel S Ointment | Traumeel S Gel | Diclofenac Gel | Total
Number analyzed (Participants) | 143 | 140 | 137 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 143 | 140 | 137 | 420
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 34 | 112
  Male | 104 | 101 | 103 | 308
Region of Enrollment [Number; unit: participants]
  Spain | 143 | 140 | 137 | 420

OUTCOME MEASURES:

1. Primary Outcome: Patient's Assessment of Ankle Pain (VAS)- Absolute Value Decrease on Day 7
Description: Pain evaluated by a 100 mm visual analogue scale (VAS) where 0 means no pain and 100 means the highest, unbearable pain. The absolute values of VAS have been the basis of analysis.
  The highest is the change in negative, the better are the results in absolute values.
Time Frame: From baseline (day 1) visit to day 7
Population: Changes from baseline at day7: absolute values and in percentage. Primary analyses were based on the Intent-To-Treat sample. Only patients with intial VAS<30 mm were excluded from the analysis set. Missing data were handled by the 'Last Observation Carried Forward' method.
Measure: Median (Inter-Quartile Range); unit: Absolute value units on a scale VAS
Arm/Group | Traumeel S Ointment | Traumeel S Gel | Diclofenac Gel
Number analyzed (Participants) | 143 | 140 | 137
Absolute value units on a scale VAS | -33.00 [-45.40 to -23.70] | -37.10 [-50.00 to -27.30] | -37.10 [-47.40 to -26.80]

2. Primary Outcome: Change of the Foot and Ankle Ability Measurement (FAAM), Activity of Daily Living Subscale (ADL) From Baseline to Day 7
Description: The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: the Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale.
  Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' (score 4), ´slight difficulty´, ´moderate difficulty´, éxtreme difficulty´ to 'unable to do' (score 0). Responses marked as ´not applicable´were not counted.
  Item score totals, which range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were transformed to percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction.
Time Frame: Day 1 to day 7
Population: Changes to Baseline: absolute values. Primary analyses were based on the Intent-To-Treat sample. Only patients with intial VAS<30 mm were excluded from the analysis set. Missing data were handled by the 'Last Observation Carried Forward' method.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Traumeel S Ointment | Traumeel S Gel | Diclofenac Gel
Number analyzed (Participants) | 143 | 140 | 137
Scores on a scale | 26.20 [16.70 to 35.70] | 26.20 [16.70 to 36.90] | 25.00 [14.60 to 34.50]

3. Secondary Outcome: FAAM ADL Subscale
Time Frame: Day 1 to 4, 14, 42
Reporting Status: Not Posted

4. Secondary Outcome: FAAM Sports Subscale
Time Frame: Day 1 to 4, 7, 14, 42
Reporting Status: Not Posted

5. Secondary Outcome: Swelling ('Figure-of-eight')
Time Frame: Day 1 to 4,7,14
Reporting Status: Not Posted

6. Secondary Outcome: Physician's Assessment of Normal Function/Activity (5-point-scale)
Time Frame: Day 1 to 4, 7, 14, 42
Reporting Status: Not Posted

7. Secondary Outcome: Time to Normal Function (Training/Sports)
Time Frame: Day 1 to 4, 7, 14, 42
Reporting Status: Not Posted

8. Secondary Outcome: Global Judgment of Efficacy
Time Frame: Day 14
Reporting Status: Not Posted

9. Primary Outcome: Patient's Assessment of Ankle Pain (VAS)- Percentage Decrease on Day 7
Description: Pain evaluated by a 100 mm visual analogue scale (VAS) where 0 means no pain and 100 means the highest, unbearable pain. The absolute values of VAS have been the basis of analysis.
  The highest is the change in negative, the better are the results in percentages.
Time Frame: From baseline (day 1) visit to day 7
Measure: Median (Inter-Quartile Range); unit: Percentage change in scale VAS
Arm/Group | Traumeel S Ointment | Traumeel S Gel | Diclofenac Gel
Number analyzed (Participants) | 143 | 140 | 137
Percentage change in scale VAS | -60.55 [-85.70 to -42.90] | -71.10 [-84.85 to -48.40] | -68.90 [-83.60 to -48.95]

ADVERSE EVENTS:
Time Frame: Safety information was collected for the whole duration of the trial from 24.08.2009 (FPI) to 12.09.2011 (LPO)
Arm/Group | Traumeel S Ointment | Traumeel S Gel | Diclofenac Gel
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/148 | 0/147
Other Adverse Events (participants affected / at risk) | 11/152 | 15/148 | 8/147
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traumeel S Ointment (N=152) | Traumeel S Gel (N=148) | Diclofenac Gel (N=147)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharingitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (7) | 5 (5) | 1 (1)
Hypoasthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharingeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less